CLINICAL TRIAL: NCT01898520
Title: The Efficacy, Safety and Tolerability of Sativex as an Adjunctive Treatment to Existing Anti-spasticity Medications in Children Aged 8 to 18 Years With Spasticity Due to Cerebral Palsy or Traumatic Central Nervous System Injury Who Have Not Responded Adequately to Their Existing Anti-spasticity Medications: a Parallel Group Randomised, Double-blind, Placebo-controlled Study Followed by a 24-week Open Label Extension Phase
Brief Title: A Safety, Efficacy and Tolerability Study of Sativex for the Treatment of Spasticity in Children Aged 8 to 18 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GWSP08258
Record Dates: First submitted 2013-07-10; First posted 2013-07-12 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Cerebral Palsy
Keywords: Spasticity
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sativex (Active Comparator): Oromucosal spray containing delta-9-tetrahydrocannabinol (THC) (27 mg/mL):cannabidiol (CBD) (25 mg/mL). Each 100 μL spray to the sub-lingual or oral mucosa delivered THC 2.7 mg and CBD 2.5 mg. The maximum number of daily sprays was 12.
  Interventions: Drug: Sativex
- Placebo (Placebo Comparator): Oromucosal spray containing ethanol: propylene glycol (50:50) excipients, with peppermint oil (0.05%) flavouring and colourings FD&C Yellow No.5 (E102 tartrazine) (0.0260%), FD&C Yellow No.6 (E110 sunset yellow) (0.0038%), FD&C Red No. 40 (E129 Allura red AC) (0.00330%) and FD&C Blue No.1 (E133 Brilliant blue FCF) (0.00058%). Each 100 μL spray administered to the sub-lingual or oral mucosa delivered the colourants plus excipients. The maximum number of daily sprays was 12.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sativex — Oromucosal spray containing THC (27 mg/mL):CBD (25 mg/mL), in ethanol: propylene glycol (50:50) excipients, with peppermint oil (0.05%) flavouring. Each 100 μL spray delivered THC 2.7 mg and CBD 2.5 mg. The maximum number of daily sprays was 12.
  Other Names: Nabiximols; THC:CBD spray; GW-1000-02
  Arms: Sativex
Drug: Placebo — Oromucosal spray containing ethanol: propylene glycol(50:50) excipients, with peppermint oil (0.05%) flavouring and colourings FD&C Yellow No.5 (E102 tartrazine) (0.0260%), FD&C Yellow No.6 (E110 sunset yellow) (0.0038%), FD&C Red No. 40 (E129 Allura red AC) (0.00330%) and FD&C Blue No.1 (E133 Brilliant blue FCF) (0.00058%). Each 100 μL spray administered to the sub-lingual or oral mucosa delivered the colourants plus excipients. The maximum daily dose was 12 sprays per day.
  Other Names: GW-4000-01
  Arms: Placebo

SUMMARY:
A study to assess the effects of Sativex treatment on spasticity in a population of children and adolescents aged from 8 to 18 years with cerebral palsy or traumatic central nervous system injury. Efficacy (ability to improve symptoms), safety and tolerability will be monitored.

DETAILED DESCRIPTION:
A 12 week randomised, double-blind, placebo-controlled,parallel group study followed by a 24-week open-label extension phase.

The primary objective is to assess the efficacy of Sativex treatment using a spasticity 0-10 numerical rating scale (NRS). The endpoint for analysis is the comparison between Sativex and placebo in the change from baseline to the end of the acute phase in mean spasticity 0-10 NRS scores (week 12 or last seven days prior to withdrawal).

The secondary objectives are to assess the safety and tolerability of Sativex via volunteered adverse events, laboratory parameters and vital signs. The efficacy of Sativex compared to placebo is also investigated for the following outcomes: spasticity (modified tardieu scale (MTS) score of the most affected limb and the modified ashworth scale (MAS) score of the main muscle groups of the upper and lower limb), sleep quality (sleep 0-10 NRS), pain (paediatric pain profile [PPP]), quality of life (of both the participant and the caregiver; cerebral palsy quality of life (QOL) questionnaire and caregiver QOL questionnaire), comfort (comfort questionnaire), depression assessment (childrens depression inventory (CDI 2)) and the caregiver's global impression of change (CGIC).

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged between 8 and 18 years suffering from cerebral palsy or traumatic central nervous system injury.
* Participant and/or authorised representative willing and able to give informed consent for participation in the study.
* To have been under treatment for their spasticity for at least one year and to have reached a stage of non-progressive spasticity.
* Participant able (in the investigators opinion) and willing to comply with all study requirements.
* Participant has received inadequate efficacy and/or experienced unacceptable side effects from previous or current treatment with at least one of the following medications for spasticity:

Baclofen, Diazepam (or another benzodiazepine), Dantrolene, Tizanidine, Gabapentin, Trihexyphenidyl.

* Gross Motor Function Classification Scale Level III - V.
* MAS of two or higher in at least one muscle group.
* Participant and/or authorised representative willing for his or her name to be notified to the responsible authorities for participation in this study, as applicable in individual countries.
* Participant and/or authorised representative willing to allow his or her primary care practitioner and consultant, if appropriate, to be notified of participation in the study.

Exclusion Criteria:

* Any known or suspected history of:

  * Schizophrenia or other psychotic illness, or diagnosis of schizophrenia in a first-degree relative.
  * Alcohol or substance abuse.
* Any known or suspected hypersensitivity to cannabinoids or any of the excipients of the IMP(s)
* Use of cannabis or cannabinoid based medications (including within 30 days or 60 days of study entry respectively).
* Weight less than 15 kg.
* Female participants of child bearing potential and male participants whose partner is of child bearing potential, unless willing to ensure that they or their partner use effective contraception during the study and for three months thereafter.
* Female participant who is pregnant, lactating or planning pregnancy during the course of the study and for three months thereafter.
* Participants who have received an Investigational Medicinal Product (IMP) within the 12 weeks prior to the screening visit.
* Has been treated with botulinum toxin in the previous 12 weeks.
* Concomitant use of botulinum toxin
* Any other significant disease or disorder, which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, may influence the result of the study, or the participant's ability to participate in the study.
* Following a physical examination, the participant has any abnormalities that, in the opinion of the investigator would prevent the participant from safe participation in the study.
* Significant cardiac, renal or hepatic disease.
* Planned surgical procedure during the randomised phase of the study.
* Travel outside the country of residence planned during the study.
* Participants previously randomised into this study.
* Unwilling to abstain from donation of blood during the study

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline to the end of 12 weeks' treatment in mean spasticity 0-10 NRS score | Day 0 - Day 84
  The spasticity 0-10 NRS was completed daily at bedtime using a paper study diary. The difference between spasticity and spasm was clearly explained to the caregiver. The primary caregiver was asked the following question: "This question is about your child's muscles and how soft or tight/hard they have felt today. Think carefully about how your child's muscles have felt today and circle a number from 0 to 10 that best describes this, where: 0 = 'my child's muscles have felt totally relaxed' and 10 = 'my child's muscles have felt the tightest/hardest they have ever felt'". A reduction in score indicates an improvement in condition.
  The mean spasticity 0-10 NRS score of the last 7 days of the baseline period was used for a patient's mean baseline score. The mean 0-10 NRS score of the last 7 days prior to completion/withdrawal was used for a patient's mean end of treatment score.

SECONDARY OUTCOMES:
Change from baseline to the end of 12 weeks' treatment in mean MTS score of the most affected limb | Day 0 - Day 84
  This study looked at the MTS in the worst affected limb only. The same limb was assessed at each visit, preferably also by the same examiner.
  The MTS used the following criteria:
  * Individuals were positioned in the sitting position to test the upper extremities and a supine position to test the lower extremities
  * Three speed definitions:
    * V1 is slow as possible
    * V2 speed of limb falling under gravity
    * V3 moving as fast as possible
  * The MTS describes R1 and R2. R1 is the angle of muscle reaction; R2 is the full passive range of movement.
  * R2 is measured at V1 and R1 at V3. R2-R1 = dynamic tone component of the muscle. The relationship between R1 and R2 estimates the relative contributions of spasticity compared to contracture.
  A reduction in score indicates and improvement in condition.
Change from baseline to the end of 12 weeks' treatment in mean MAS score of the main muscle groups of the upper and lower limb | Day 0 - Day 84
  Participants were tested in the supine position and participants were instructed to relax. Muscle groups in the ankle, knee, hip, shoulder, elbow and wrist were rated on a scale of 0 = No increase in muscle tone, 1 = Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension, 1+ = Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the range of movement (ROM), 2 = More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved, 3 = Considerable increase in muscle tone, passive movement difficult, 4 = Affected part(s) rigid in flexion or extension. The MAS was performed by the same examiner at each visit, where possible. A reduction in score indicates an improvement in condition.
Change from baseline to the end of 12 weeks' treatment in mean sleep quality 0-10 NRS score | Day 0 - Day 84
  The sleep quality 0-10 NRS was completed at the same time each day, ideally when waking in the morning. This questionnaire was designed to record the level of sleep disturbance. The primary caregiver was asked the following question: "This question is about how badly your child slept last night. Please mark a number from 0 to 10 that indicates how bad your child's sleep was where: 0 = My child had a night of non-stop sleep and 10 = My child was unable to sleep at all". A reduction in score indicates and improvement in condition.
Change from baseline to the end of 12 weeks' treatment in mean Paediatric Pain Profile (PPP) score | Day 0 - Day 84
  The PPP is a 20-item behaviour rating scale designed to assess pain in children with severe neurological disability. Each item is scored on a four point scale of 0 to 3 as occurring 'not at all' (zero) to 'a great deal' (three) in the given time period. The total score therefore will range from 0 to 60. The questionnaire was designed to be completed by the child's primary caregiver and was completed at each assessment visit during the study. A reduction in score indicates an improvement in condition.
Change from baseline to the end of 12 weeks' treatment in mean cerebral palsy QOL score | Day 0 - Day 84
  The cerebral palsy QOL-Child QoL questionnaire (aged 4-12 years) is a 66-item questionnaire that looks at eight important domains of life including friends and family; participation; communication; health; special equipment; pain and bother; access to services; and parents' health. Completed by the primary caregiver it assesses how the caregiver thinks the child feels about these aspects of their life. The numbers range from one (very unhappy) to nine (very happy).
  The teen questionnaire (aged 13-18 years) comes with two questionnaires, one to be completed by the participant, if applicable, and one by the primary caregiver. The first seven sections of the questionnaire are identical and look at seven important domains of life including friends and family; school; participation; communication; health, special equipment and pain and bother. The caregiver questionnaire has an additional section which looks at access to services.
  Increases in score indicate an improvement in condition.
Change from baseline to the end of 12 weeks' treatment in mean comfort questionnaire outcome (time spent sitting in comfort) | Day 0 - Day 84
  The comfort questionnaire was completed at the same time each day, i.e. bedtime in the evening. The caregiver was asked to reflect on the whole day and record the longest number of minutes at any one time over which their child was able to sit in comfort for, without moving position. An increase in time indicates an improvement in condition.
Change from baseline to the end of 12 weeks' treatment in mean CDI 2 score | Day 0 - Day 84
  The CDI 2 contains 28 items, each of which consists of three statements (each scored 0-2 [0=best outcome, 2=worst outcome]). For each item, the participant is asked to select the statement that best describes his or her feelings. The assessment is designed for a variety of situations, including schools, child guidance clinics, pediatric practices, and child psychiatric settings. If the participant is unable to complete the questionnaire, the questionnaire will be left blank.
  A reduction in score indicates an improvement in condition.
Change from baseline to the end of 12 weeks' treatment in mean caregiver QOL (SF-36-II) score | Day 0 - Day 84
  The SF-36-II is a 36 item questionnaire that measures eight multi-item dimensions of health: physical functioning (10 items) social functioning (two items) role limitations due to physical problems (four items), role limitations due to emotional problems (three items), mental health (five items), energy/vitality (four items), pain (two items), and general health perception (five items). There is a further unscaled single item asking respondents about health change over the past year. For each dimension item scores are coded, summed, and transformed on to a scale from 0 (worst possible health state measured by the questionnaire) to 100 (best possible health state). An increase in score indicates an improvement in condition.
CGIC response on participants general functional capabilities at the end of 12 weeks' treatment | Day 84
  The main caregiver was asked to assess the change in the participant's condition. Questions were rated on a seven-point scale: Very much worse, Much worse, Minimally worse, No change, Minimally better, Much better, Very much better. The caregiver was asked:
  "How have the participant's general functional abilities changed since Visit 2?" (i.e. change from baseline).
  The number of participants for each marker is presented.
CGIC response on participants ease of transfer at the end of 12 weeks' treatment | Day 84
  The main caregiver was asked to assess the change in the participant's condition. Questions were rated on a seven-point scale: Very much worse, Much worse, Minimally worse, No change, Minimally better, Much better, Very much better. The caregiver was asked:
  "How has the participant's ease of transfer changed since Visit 2?"(i.e. change from baseline).
  The number of participants for each marker is presented.
The incidence of adverse events during the randomised treatment period | Day 0 - Day 84
  The number of participants who reported an adverse event during the randomised treatment part of the study is presented.

CONTACTS AND LOCATIONS:
Locations (14):
- Center 14, Prague, Czechia
- Israel (2):
  - Center 7, Tel Aviv
  - Center 8, Tel Litwinsky
- United Kingdom (11):
  - Center 2, Bristol
  - Center 6, Cambridge
  - Center 10, Exeter
  - Center 13, Glasgow
  - Center 3, Liverpool
  - Center 1, London
  - Center 5, London
  - Center 12, Norwich
  - Center 9, Nottingham
  - Center 11, Salisbury
  - Center 4, Sheffield